CLINICAL TRIAL: NCT06154564
Title: PAMNEU: Easy Detection of Memory Disorders Using Very Short ALBA and PICNIR Tests in Neurological Outpatient Clinics in the Czech Republic
Brief Title: PAMNEU - Memory in Neurology
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Tadeáš Mareš, Consultation-liaison psychiatrist, Charles University, Czech Republic
Other Study IDs: PAMNEU
Record Dates: First submitted 2023-11-19; First posted 2023-12-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment
Keywords: Cognitive Impairment; Outpatient Neurologic Service; Population Distribution
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observed group: No intervention will be administered on behalf of the project. The participants will be tested using ALBA and PICNIR (non-invasive) cognitive tests, and further FAQ-CZ and GDS-CZ questionnaires will be administered.

SUMMARY:
Memory in Neurology project (PAMNEU) aims to map the distribution and severity of cognitive impairment in patients of outpatient neurologic offices across the geographical area of the Czech Republic. 1000 patients in 50 neurologic offices will undergo cognitive tests (ALBA and PICNIR) and psychometric scales (FAQ-CZ and GDS-CZ) to asses their functional state and depressive symptoms.

The trial's primary goal is to assess the distribution of cognitive impairment among diagnostic groups in neurologic care according to the ICD-10. Additionally, the feasibility of ALBA and PICNIR methods to uncover previously undiagnosed cognitive impairments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Dispensarization of at least six months in an outpatient neurologic office with an ICD-10 diagnosis
* Age>=50
* Permanent residency in the geographical area of the Czech Republic

Exclusion Criteria:

* Diagnosis of mental retardation (F70-F79) according to ICD-10
* Refusal to sign the informed consent and consent with GDPR
* Uncorrected visual impairment
* Uncorrected auditory impairment
* Impairment of hand movement preventing the patient from filling in the questionnaires.
* Inability to participate in the project

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is intended to be comprised of persons (50yrs+) living in the geographical area of the Czech Republic undergoing treatment at an outpatient neurologic office for a diagnosis defined in ICD-10 (excluding mental retardation). The probability sample will be created by a random selection of persons undergoing their regular outpatient neurologic checkups.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Baseline ALBA | Established on Day 0 as a single assessment.
  Amnesia Light and Brief Assessment (ALBA) test is an innovative method to assess cognitive functions quickly. The cognitive performance is scaled as an overall score between 0-12 (a lower value denotes a more severe cognitive impairment).
Baseline PICNIR | Established on Day 0 as a single assessment.
  Picture Naming and Immediate Recall test (PICNIR) is an innovative test method to assess cognitive functions quickly. The cognitive performance is scaled as an overall score between 0-20 (a lower value denotes a more severe cognitive impairment).
Statistical analysis of ALBA results | The final statistical analysis will be performed through study completion, an average of 6 months.
  Statistical analysis of ALBA results compared to groups determined by ICD-10 diagnosis and demographical data.
Statistical analysis of PICNIR results | The final statistical analysis will be performed through study completion, an average of 6 months.
  Statistical analysis of PICNIR results compared to groups determined by ICD-10 diagnosis and demographical data.

SECONDARY OUTCOMES:
Baseline FAQ-CZ | Established as a baseline on Day 0.
  Functional Activities Questionnaire - Czech version (FAQ-CZ) is a standardized questionnaire administered to assess a patient´s functional state regarding daily activities. Ten items of daily functioning are scaled between 0-3 (a higher value denotes a higher dependency) to reach the overall score between 0-30 (a higher value denotes a higher dependency). This version of the scale will be used for participants´ self-evaluation.
Baseline GDS-CZ | Established as a baseline on Day 0.
  The Geriatric Depression Scale - Czech version (GDS-CZ) is a standardized questionnaire administered to assess depressive symptoms, particularly in the elderly population. Fifteen items are scaled between 0-1 to reach the overall score between 0-15 (a higher value denotes a higher level of depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Aleš Bartoš, M.D., Ph.D., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Teaching Hospital Královské Vinohrady, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD is to be shared upon request by a verified researcher. The study director´s discretion is reserved.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon the final publication of the outcomes, indefinitely.
Access Criteria: Being a verified researcher.